CLINICAL TRIAL: NCT06099119
Title: Open Label Randomized, Multicentre, Controlled Trial of Pancreatic Enzyme Replacement Therapy (PERT) for Pancreatic Exocrine Insufficiency (PEI) in Patients With Unresectable Pancreatic Cancer. The PERTseverance Trial.
Brief Title: Efficacy of PERT for PEI in Unresectable Pancreatic Cancer.
Acronym: PERTseverance
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Complejo Hospitalario de Navarra (Other); Karolinska Institutet (Other); San Raffaele University Hospital, Italy (Other); Beaujon Hospital (Other)
Responsible Party: Principal Investigator, J. Enrique Domínguez-Muñoz, Prof. PhD. MD., Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEI004/2021
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental arm (Experimental): Creon 35.000 Ph.U (R) at a fixed dose of 3 capsules orally with main meals (breakfast, lunch and dinner) and 2 capsules with snacks over 6 months post randomization.
  Interventions: Drug: creon 35.000 Ph.U (R)
- control arm (Other): Creon 35.000 Ph.U (R) at a fixed dose of 3 capsules orally with main meals (breakfast, lunch and dinner) and 2 capsules with snacks during the last 3 months post randomization.
  Interventions: Other: Best Standarard of Care

INTERVENTIONS:
Drug: creon 35.000 Ph.U (R) — Experimental arm: Pancreatic Exocrine Replacement Therapy (PERT) treatment during the six months study period.
  Arms: experimental arm
Other: Best Standarard of Care — Control arm: no treatment over 3 months from randomization. PERT from third month untill last visit in sixt month
  Other Names: creon 35.000 Ph.U (R)
  Arms: control arm

SUMMARY:
- This will a be an open label, multicentre, randomized, controlled study in patients with unresectable pancreatic cancer, locally advanced or metastatic, with significant weight loss, and the tumour located in the head of the pancreas associated with dilated main pancreatic duct. Pancreatic Exocrine Replacement Therapy (PERT) in these patients will be given on top of other required therapies (best standard of care, BSC), including oncologic therapies, diabetes mellitus therapies and acid suppressants and nutritional support as appropriate. The duration of the study will be up to six months.

Consecutive patients meeting inclusion criteria and none of the exclusion criteria will be evaluated for the study. Those patients signing the informed consent for study participation will be randomized to one of the following two arms:

* The experimental arm will receive the best standard of care (BSC) and PERT (capsules containing pancreatin 35,000 Ph.U.) at a fixed dose of 3 capsules with main meals (breakfast, lunch and dinner) and 2 capsules with snacks over 6 months.
* The control arm will receive the BSC over 3 months, followed by a further 3-month open uncontrolled phase of BSC + PERT at the dose mentioned above.

All patients will receive in addition a proton pump inhibitor (PPI) bid (any PPI at standard dose is acceptable -omeprazole 20 mg, lansoprazole 30 mg, pantoprazole 40 mg, rabeprazole 20 mg, esomeprazole 40 mg) while on PERT, 20-30 minutes before breakfast and dinner.

To make the two arms comparable, patients will be stratified in two groups (locally advanced and metastatic pancreatic cancer) for randomization using computer generated random numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed unresectable, locally advanced or metastatic, pancreatic cancer.
2. Tumour located in the head of the pancreas.
3. Dilated main pancreatic duct confirmed by imaging methods (CT scan, MRI and/or EUS).
4. Significant weight loss (≥5% of the usual body weight) at screening.
5. Life expectancy of at least six months at screening.
6. Signed informed consent to the study.

Exclusion Criteria:

1. Hypersensitivity to pancreatin of porcine origin or to any of the excipients.
2. Patients on neoadjuvant therapy, or in whom neoadjuvant therapy is planned.
3. Patients already on PERT.
4. Prior history of upper gastrointestinal or pancreatic surgery.
5. Short life expectancy (shorter than 6 months).
6. Patients on second line or beyond chemotherapy (those who failed with first line chemotherapy therapy).
7. Patients in whom a pancreatic stent has been placed.
8. Unsolved gastric outlet obstruction.
9. Unwillingness to participate in the study.
10. Inability to comply with the study visits and study protocol, whatever the reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight over study period. | From visit 1 day 1 to visit 4 sixt month.
  ƍ between visit 4 (sixt month) and visit 1 (day 1) in the patient's weight

CONTACTS AND LOCATIONS:
Locations (4):
- Istituto di Ricovero e Cura Carattere Scientifico San Raffaele, Milan, Milan, Italy
- Spain (2):
  - University Hospital of Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario de Navarra, Pamplona, Navarre
- Karolinska Institutet, Stockholm, Stockholm County, Sweden